CLINICAL TRIAL: NCT02219529
Title: Magnetic-controlled Capsule Endoscopy vs. Gastroscopy for Detection of Gastric Diseases: A Prospective Self-controlled Comparative Multicenter Trial
Brief Title: Magnetic-controlled Capsule Endoscopy vs. Gastroscopy for Detection of Gastric Diseases
Acronym: MCE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Changhai Hospital (Other)
Collaborators: RenJi Hospital (Other); Nanfang Hospital, Southern Medical University (Other); Chinese PLA General Hospital (Other); General Hospital of Beijing PLA Military Region (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Shandong Provincial Hospital (Other Government); Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Director of Gastroenterology Dept., Changhai Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: MCE-1
Record Dates: First submitted 2014-08-12; First posted 2014-08-19 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Gastric Diseases,; Gastric Ulcer,; Gastric Polyps,; Early Gastric Cancer,; Chronic Gastritis
MeSH Terms: conditions — Stomach Diseases; Stomach Ulcer; Polyposis, Gastric; Stomach Neoplasms | interventions — Endoscopy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MCE (Experimental): patients were assigned to swallow MCE first, followed by the gastroscopy
  Interventions: Device: MCE
- Standard gastroscopy (Active Comparator): patients were assigned to swallow MCE first, followed by the gastroscopy
  Interventions: Device: Standard gastroscopy

INTERVENTIONS:
Device: MCE
  Other Names: magnetic-controlled capsule endoscopy
  Arms: MCE
Device: Standard gastroscopy
  Arms: Standard gastroscopy

SUMMARY:
A new Magnetic-controlled Capsule Endoscopy (MCE) was developed by ANKON and got SFDA's approval in China in 2013. It has recently been evaluated to compare the diagnostic accuracy of MCE with that of standard gastroscopy for gastric diseases in 70 patients with encouraging results (In Press). To further testify the diagnostic accuracy of MCE for both the diffuse and focal diseases in stomach, we performed this single-blinded multi-center prospective study compared MCE with gastroscopy in patients with gastric symptoms and indication for upper GI Endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients presented with gastric symptoms and ready for the first Upper GI endoscopy
* Patients with known focal gastric diseases: gastric ulcer, gastric polyps, early gastric cancer, gastric stromal tumors and so on.
* Age of 18 years to 70 years

Exclusion Criteria:

* Patients with impaired bowel movement from ileus or organic digestive diseases
* Patients with known large and obstructing tumors of the upper GI tract
* Patients after upper GI surgery or abdominal surgery altering GI anatomy
* Patients under full anticoagulation
* Patient in poor general condition
* Patients using equipment that may be affected by radio transmission
* Patients using equipment that may be affected by magnetic field
* Pregnancy or suspected pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2014-08; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Number of subjects diagnosed with gastric diffuse lesions by MCE Versus Standard Gastroscopy | 2 days
Number of gastric focal lesions founded by MCE Versus Standard Gastroscopy | 2 days

SECONDARY OUTCOMES:
Volume of water and drugs used for gastric preparation | 1 hour
Scores of the cleanliness of stomach after preparation | 1 day
Percentage of patients in whom there was complete visualization of the gastric surface in the antrum, body, and fundus and identification of the cardia and pylorus | 1 day
Examination times of MCE and standard gastroscopy | 1 day
Patient acceptance of MCE and standard gastroscopy | 3 days
Adverse events of both procedures | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoshen Li, Prof., Principal Investigator — Changhai Hospital
Locations (1):
- Shanghai Changhai Hospital, Shanghai, China

REFERENCES:
- [Background] Liao Z, Duan XD, Xin L, Bo LM, Wang XH, Xiao GH, Hu LH, Zhuang SL, Li ZS. Feasibility and safety of magnetic-controlled capsule endoscopy system in examination of human stomach: a pilot study in healthy volunteers. J Interv Gastroenterol. 2012 Oct-Dec;2(4):155-160. doi: 10.4161/jig.23751. Epub 2012 Oct 1. PMID 23687601
- [Background] Liao Z, Gao R, Xu C, Li ZS. Indications and detection, completion, and retention rates of small-bowel capsule endoscopy: a systematic review. Gastrointest Endosc. 2010 Feb;71(2):280-6. doi: 10.1016/j.gie.2009.09.031. PMID 20152309
- [Derived] Liao Z, Hou X, Lin-Hu EQ, Sheng JQ, Ge ZZ, Jiang B, Hou XH, Liu JY, Li Z, Huang QY, Zhao XJ, Li N, Gao YJ, Zhang Y, Zhou JQ, Wang XY, Liu J, Xie XP, Yang CM, Liu HL, Sun XT, Zou WB, Li ZS. Accuracy of Magnetically Controlled Capsule Endoscopy, Compared With Conventional Gastroscopy, in Detection of Gastric Diseases. Clin Gastroenterol Hepatol. 2016 Sep;14(9):1266-1273.e1. doi: 10.1016/j.cgh.2016.05.013. Epub 2016 May 20. PMID 27211503
- See also: Related Info — http://www.csde.org.cn/